CLINICAL TRIAL: NCT05695846
Title: Development of Physiology- and Pathophysiology-based Diagnostic Tests and Therapeutics for Patients With Pharyngeal Reflux of Gastric Content
Brief Title: Diagnostic Tests in Supra-Esophageal Gastroesophageal Reflux Disease (SE-GERD)
Acronym: SE-GERD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty in recruiting subjects led to no enrolment in the protocol.
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Reza Shaker, MD, Associate Provost for Clinical and Translational Research, Senior Associate Dean and Director of the Clinical and Translational Science Institute of SE WI, and the Joseph E. Geenen Professor and Chief of Gastroenterology and Hepatology, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRO00020732
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: GERD patients with complaints of regurgitation and supra-esophageal symptoms
Masking Description: Data analysis staff will be blinded with regard to patient status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patients with supra-esophageal gastroesophageal reflux disease (Other): GERD patients with complaints of regurgitation and supra-esophageal symptoms
  Interventions: Device: externally applied cricoid cartilage pressure

INTERVENTIONS:
Device: externally applied cricoid cartilage pressure

SUMMARY:
After defining the manometric characteristics of UES incompetence associated with documented pharyngeal reflux, we will determine the reproducibility of manometric criteria for UES incompetence in prevention of pharyngeal reflux. We hypothesize that these criteria are comprised of either a single or constellation of manometric abnormalities. After determining the ability of externally applied cricoid cartilage pressure in preventing pharyngeal reflux, we further hypothesize that this approach will eliminate or reduce esophago-pharyngeal reflux by enhancing the UES pressure barrier. We anticipate there will be a close spatial correlation between the site of applied pressure and area of increased pressure within UES high pressure zone. Lastly, we will determine and characterize the effect of externally applied cricoid cartilage pressure on related functions such as belch and swallow, testing the hypothesis that these functions will not be impaired.

DETAILED DESCRIPTION:
Study subjects: we will study gastroesophageal reflux disease (GERD) patients with complaint of regurgitation and one of the following supra-esophageal symptoms attributed to reflux of gastric content: chronic cough, frequent throat clearing, history of non-deglutitive aspiration pneumonia, hoarse voice, chronic sinusitis and dental erosion i.e. Supraesophageal gastroesophageal reflux disease (SE-GERD). The presence of GERD will be verified in their records by result of prior endoscopy or pH monitoring within the past two years. It not, they will undergo transnasal esophagogastroduodenoscopy (T-EGD). If negative, they will undergo pH monitoring off medications to ascertain presence of GERD according to clinically accepted criteria (AGA guidelines (39). We will not enroll patients with functional heartburn (Rome III criteria (40). For Supra-esophageal complications we will use the endoscopic criteria used in clinical Ear, Nose and Throat (ENT) practice and validated symptom severity index questionnaire (developed by Belafsky et al) with the help of our otolaryngologist co-investigator Dr. Joel Blumin.

Study position: studies will be done in supine postures due to vulnerability of the airway in this position.

Instrumentation: all instrumentations will be trans-nasal following application of 2% lidocaine limited to the nasal cavity.

Study technique: concurrent video-pharyngo-laryngoscopy and combined high-resolution manometry and impedance recording along with pH monitoring.

All study participants will give written informed consent followed by filling out a general health questionnaire. Additionally, a Belafsky Index will also be filled out in the same session by the study participant to assess the level of symptoms within the last month associated with supraesophageal reflux.

Combined manometric/impedance/pH recording: we will use combined solid-state high resolution manometry and impedance catheter with 36 circumferential pressure sensors, spaced 1 cm apart (Sierra Scientific, Los Angeles, CA) 18 impedance sensor couplets spaced 2 cm apart measuring at a sample rate of 40 Hz (Given Imaging Duluth, GA), 3 pH sensors spaced 7 and 10 cm respectively. The catheter will be introduced transnasally in a fashion that at least 3 proximal manometric sensors are in the pharynx and two impedance and one pH sensors are located 2 cm proximal to upper margin of UES in the pharynx. With this arrangement 3-4 manometric and one or two impedance couplets will be positioned in the UES high pressure zone while the remaining pressure sensors will cover the sub-sphincteric striated segment and the rest of esophagus along with lower esophageal sphincter (LES) through very proximal portion of stomach, although in very tall participants the full length of LES may not be covered. One ph sensor will be 3cm distal to UES while the remaining impedance couplets will span the proximal and distal esophagus.

Concurrent videopharyngo-laryngoscopy: to monitor concurrently the pharynx and larynx for entry of simulated refluxate we will use a Pentax FNL-10AP laryngopharyngoscope passed through the other nostril and positioned within the pharynx such that the UES inlet, vocal cords and pyriform sinuses are visualized. The laryngopharyngoscopic images will be synchronized with manometric/impedance/pH recordings by importing and superimposing the endoscopic images onto high resolution manometric recordings. Using a specially designed timer (Thalner Electronics Labs, Inc, Ann Arbor, MI) time in hundredths of a second will be superimposed on the video images for durational analyses of endoscopic images.

Slow and rapid intraesophageal infusion: A 3 mm outer diameter injection tube will be placed through the same nostril in a fashion that the injection port will be located 5-7cm above the manometrically determined upper border of lower esophageal sphincter (LES). With this arrangement gastroesophageal reflux events will be simulated by intra-esophageal injection of body temperature infusates namely,1/2 normal saline (its ionic nature helps impedance recording and identification of intra-esophageal distribution), 0.1 N HCl. As stated above infusions will be done in three sessions. Slow acid and slow1/2saline sessions will test two volumes (20 and 60ml) and two rates (.05 and 1.0 ml pre second). Since our preliminary data suggest a strong differentiating capacity for slow infusion (1ml/sec) in uncovering UES abnormalities we propose to test two slow infusions to identify the one with most differentiating capacity. We study slow acid and saline perfusion in two sessions to avoid the issue of esophageal sensitization effect on saline distension in addition to reasons describe above. The rapid injection session will test two volumes (20 and 60 ml) and one rate (10 ml per second). In this session we will test both acid and saline due to short contact time of the acid which make the sensitization less likely. A modified Harvard pump will be used for infusions. Each infusion will be repeated three times. The order of infused material as well as the volume of infused material in all sessions will be randomized. Also randomized, will be the three different study sessions. Liquid infusates will be colored green using food dye for ease of recognition of pharyngeal reflux. Exact timing and type of the injection will be documented using the event marker feature of the Manoscan® system. Each perfusion will be performed only when the UES, esophagus and LES are at baseline for at least three tidal volume respiratory cycles and 20s after a preceding peristaltic event. After each perfusion, manometry will be carefully monitored for 20s and then subjects will be cued to swallow and clear their esophageal contents. Esophageal clearance will be verified by the presence of an effective peristalsis and return of intra-esophageal impedance and pressure to baseline. As stated above infusions will be done in three sessions within the same two hour study visit.. Endoscopic views of pharynx will be watched carefully during infusions. At the first sign of reflux, perfusion will be stopped and participants will be instructed to swallow to avoid any potential airway compromise. This technique has been used in our laboratory for the past three years without any problem.

Pressure Data Analysis: All pressure measurements will be recorded at a 35HZ frequency and measured in reference to the atmospheric pressure UES and LES pressures will be measured utilizing the e-sleeve function of the Manoview ® software. All UES, LES and esophageal baseline pressures will be measured as peaks and troughs over 3 tidal volume respiratory cycles at stable resting conditions when no pharyngeal, gastric, esophageal, UES or LES events are present. Type, frequency, amplitude, onset, and duration of the UES response along with the LES and esophageal body response will be recorded.

UES pressure response to intraesophageal infusion: Percent UES relaxation and percent UES contraction will be calculated as a fraction of the maximum possible relaxation (baseline UES pressure-proximal esophageal pressure) and as a fraction of the maximum UES contraction pressure, respectively. UES relaxation will be considered complete (100%) if an audible belch is documented or the nadir UES pressure at least equalizes to the proximal esophageal pressure. Due to considerable variability of the resting UES pressure even at rest we have set a conservative threshold (10 mmHg) for determining the UES response (43-44). UES response will be categorized as an ordinal variable: contraction (UES pressure exceeds the peak baseline pressure by more than 10 mmHg); relaxation (UES pressure drops more than 10 mmHg below baseline trough pressure); or no response. It has been observed that often prior to and almost always after a swallow related UES relaxation (as UES participates in pharyngoesophageal peristaltic wave) there is an increase in UES tone that has been linked to the preceding relaxation rather than an independent event therefore, we will consider the UES contraction as a response only if it is not preceded by a UES relaxation response and not followed by UES relaxation within 3 seconds.

Extent of esophageal intraluminal pressure increase during infusions: will be recorded as an ordinal variable: 1) if esophageal pressure increase more than 3 mmHg above baseline during perfusion, esophageal pressure and peak rate of pressure increase (dp/dt) within a 0.1 s window will be measured during the perfusion in the proximal and distal esophageal segments as continuous variables.

Esophageal clearing response to intra-esophageal perfusion: will be classified into four categories: 1/ simultaneous esophageal contraction (>20 mmHg); 2/ secondary peristalsis as a sequential esophageal contraction of at least 5cm length and amplitude greater than 20 mmHg without preceding swallow related pharyngeal contraction); 3/ primary peristalsis (>20 mmHg) as an orderly sequential esophageal contraction of at least 5cm length and amplitude greater than 20 mmHg preceded by pharyngeal contraction and UES relaxation ; and, 4/ no response as the esophageal body pressure changes less than 20 mmHg or 5cm length during 20 second analysis window. We will monitor clearance of the infusate from esophagus by impedance monitoring up to 60 seconds and then subjects will be instructed to swallow until esophageal contents clear.

LES response to intraesophageal perfusion: Although LES function is not the center of present proposal when available its response to infusion will be classified into three types: 1/ complete relaxation defined as equalization of the LES pressure to gastric pressure; 2/ partial relaxation defined as a pressure drop > 5 mmHg; and, 3/ no response. The predominant UES, LES and esophageal response will be considered mode of three trials and recorded as an ordinal variable.

Videoendoscopic data analysis: onset of the entry of colored refluxate into the pharynx though the UES inlet will be determined and correlated with the UES, esophageal and LES pressure phenomena, impedance and pH events. Endoscopic documentation of pharyngeal reflux will be considered the gold standard and impedance and pH data will be compared to it.

Identification of biologic events: Glottal kinetics and movements as well as changes in the geometry of pharyngeal cavity will be used to identify swallow esophago-glottal closure reflex and belch. Belch and swallow will also be identified by their characteristic pressure and impedance signatures, investigator observation and participant signaling using a marker and correlated with endoscopic findings for certainty.

Criteria for abnormal UES barrier function: Based on our preliminary data these include, presence of one or any constellation of the following: absence of sustained UES contraction, transient partial or complete relaxation. Additional criteria may include absence of striated esophagus peristalsis or absence of secondary peristalsis. Presence of simultaneous contraction or lack any contraction. These criteria will be applied to infusion period (60 sec) plus two minute post-infusion.

Criteria for normal UES barrier function: sustained contraction of at least 20mmHg above pre-infusion period (three respiratory cycles) in response to infusion for the duration of infusion and lack of the abnormal criteria stated above.

Determine the ability of externally applied cricoids cartilage pressure on preventing pharyngeal reflux: Our preliminary studies have shown that externally applied pressure on the cricoid cartilage (20mmHg) can increase the intraluminally recorded UES pressure. These studies have also shown that this technique can prevent experimentally induced pharyngeal reflux in patients with SE-GERD and regurgitation. UES high pressure zone ranges from 3-4cm and is generated by participation of inferior pharyngeal constrictor, cricopharyngeus muscle and most proximal part of the esophagus. The spatial relationship of externally applied pressure and the UES pressure profile has not been studied. It is also not known whether external pressures applied, not exactly on the cricoid could impart the same effect. Our preliminary data suggests location dependent effect on UES pressure profile. Because this approach may have practical clinical ramification, in this sub-aim, we will characterize the effect of a 20mmHg pressure, externally applied to and several points distal and proximal to the cricoid cartilage on UES pressure profile. We have chosen 20 mmHg pressure based on our preliminary data. This procedure will be performed on all EPR patients recruited into our study. Each apparatus for exerting external cricoid pressure is custom fitted for each subject at the time of the study. Furthermore, the ICF for this protocol has been edited to include this procedure in the description of test performed during each experiment

Determine and characterize the effect of externally applied cricoid cartilage pressure on related functions such as belch and swallow: We will test dry, 5 and 10 ml ½ saline swallowsX3 in random order. In addition we will test belching by injecting various volumes of air into the esophagus through the previously paced infusion catheter. We will test 20 and 40 ml room TX3. Studies will be done with and without application of cricoid pressure. Cricoid pressure will be applied at 20mmHg by using our laboratory made neck band as described above with the exception that the pressure bar will be 10X30mm to cover the width of the cricoid cartilage for maximum effect. These studies will be carried out with the test subjects in the upright and supine positions.

ELIGIBILITY:
Inclusion Criteria:

* GERD patients with complaints of regurgitation and supra-esophageal symptoms will be included Patient definition will be based on position statement and technical reviews of the American Gastroenterological Association and Montreal definition and classification of gastroesophageal and reflux disease (Am J Gastroenterol. 2006;101:1900-1920).

Exclusion Criteria:

* Age <20 or >85

  * History or active alcohol or drug abuse
  * History of upper GI and ears, nose, throat and pulmonary diseases that may affect the oropharyngoesophageal axis and stomach
  * History of malignancy and chemo-radiation therapy
  * Unable to give consent
  * Pregnant women (see justification in the Women and Minority Inclusion in Clinical Research section).
  * History of allergy to Lidocaine for nasal topical anesthesia.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01-29 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-04-02 (Actual)

PRIMARY OUTCOMES:
Endoscopic evidence of supra-esophageal reflux | Procedure (During simulated reflux perfusion of the esophagus)
  Visually confirmed supra-esophageal refluxate seen during video endoscopy and log the number of reflux episodes duing each simulated esophageal reflux infusion

CONTACTS AND LOCATIONS:
Overall Officials: Reza Shaker, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Reza Shaker, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No